CLINICAL TRIAL: NCT04262609
Title: Faecal Incontinence in Prostate Cancer Survivors Treated With Moderately Hypofractionated Radiotherapy
Brief Title: Faecal Incontinence in Prostate Cancer Survivors Treated Whith Radiotherapy
Status: Active, not recruiting | Type: Observational
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Joan Lozano Galan, Principal investigator, Consorci Sanitari de Terrassa
Other Study IDs: ONCORTCST2020-1
Record Dates: First submitted 2020-02-05; First posted 2020-02-10 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Faecal Incontinence; Prostate Cancer
Keywords: hypofractionated radiotherapy; quality of life; cancer survivors
MeSH Terms: conditions — Encopresis; Prostatic Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: hypofractionated radiotherapy — volumetric modulated moderately fractionated arc therapy

SUMMARY:
The objective of the study is to determine the incidence of faecal incontinence in prostate cancer survivors treated with moderately hypofractionated radiation therapy and correlate the dose received by the anal sphincter with the degree of faecal incontinence.

DETAILED DESCRIPTION:
The investigators know that high doses of irradiation in the anal sphincter are associated with more chronic fecal leaks in survivors irradiated by normofractionated radiotherapy prostate cancer.

The safe dose of irradiation of the anal sphincter with radiotherapy modern techniques (volumetric modulated arc therapy with moderately hypofracctionation) is unknown.

Urgency and faecal incontinence greatly affects the quality of life of these patients.

Therefore, it is interesting to implement strategies to protect the anatomical structures involved in fecal continence.

The objective of the study is to determine the incidence of faecal incontinence in prostate cancer survivors treated with modern moderately hypofractionated radiation therapy and correlate the dose received by the anal sphincter with the degree of faecal incontinence.

The investigators also want to evaluate the quality of life of these patients

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer survivors treated in our department by hypofractionated radiotherapy

Exclusion Criteria:

* Relapse of prostate cancer
* Other active cancer
* Mental disorder

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Prostate cancer survivors treated in our department by volumetric modulated hypofractionated arc therapy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
faecal incontinence after prostate radiation therapy | before radiotherapy (basal)
  grade of faecal incontinence in prostate cancer patients
faecal incontinence after prostate radiation therapy | change 2 years after completion of radiotherapy
  grade of faecal incontinence in prostate cancer survivors
faecal incontinence after prostate radiation therapy | change 3 years after completion of radiotherapy
  grade of faecal incontinence in prostate cancer survivors
faecal incontinence after prostate radiation therapy | change 4 years after completion of radiotherapy
  grade of faecal incontinence in prostate cancer survivors
faecal incontinence after prostate radiation therapy | change 5 years after completion of radiotherapy
  grade of faecal incontinence in prostate cancer survivors

SECONDARY OUTCOMES:
Quality of life after prostate radiation therapy | 3 years after completion of radiotherapy
  Quality of life in prostate cancer survivors comparing continents patients and incontinents patients
Quality of life after prostate radiation therapy | 5 years after completion of radiotherapy
  Quality of life in prostate cancer survivors comparing continents patients and incontinents patients

CONTACTS AND LOCATIONS:
Overall Officials: Joan Lozano, MD, Principal Investigator — Consorci Sanitari de Terrassa
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lozano J, Feltes N, Colomer M, Lizondo M, Carmona M, Romero C, Ribas Y, Paredes S, Galdeano M, Sole JM. Fecal incontinence after moderately hypofractionated volumetric modulated arc therapy for prostate cancer: incidence and impact on quality of life. Clin Transl Oncol. 2025 Oct;27(10):4003-4010. doi: 10.1007/s12094-025-03926-w. Epub 2025 Apr 22. PMID 40261490